CLINICAL TRIAL: NCT00054171
Title: A Pilot Study of Short (1-2.5 h), Medium (4-6 h) and Long (18-24 h) Applications of 20% Topical ALA-PDT for Photodynamic Therapy of Cutaneous T and B Cell Lymphomas and Cutaneous Infiltrates of Early CLL
Brief Title: Photodynamic Therapy in Treating Patients With Lymphoma or Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: DS 97-32; RPCI-DS-9732
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Leukemia; Lymphoma
Keywords: B-cell chronic lymphocytic leukemia; stage I cutaneous T-cell non-Hodgkin lymphoma; stage I mycosis fungoides/Sezary syndrome; stage 0 chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome | interventions — Aminolevulinic Acid

INTERVENTIONS:
Drug: aminolevulinic acid hydrochloride

SUMMARY:
RATIONALE: Photodynamic therapy uses light and drugs that make cancer cells more sensitive to light to kill cancer cells. Photosensitizing drugs such as aminolevulinic acid are absorbed by cancer cells and, when exposed to light, become active and kill the cancer cells.

PURPOSE: Randomized phase II trial to study the effectiveness of photodynamic therapy using aminolevulinic acid in treating patients who have cutaneous T-cell lymphoma, B-cell lymphoma, or early chronic lymphocytic leukemia involving the skin.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the pain grade and epidermal toxic response (ETR) of patients with T-cell or B-cell lymphoma or early chronic lymphocytic leukemia with cutaneous infiltrates treated with photodynamic therapy using aminolevulinic acid.
* Determine the feasibility of maintaining a pain grade of 1 or less and an approximate ETR of 2 in patients receiving up to 12 sessions of this regimen.
* Determine the maximal irradiance and corresponding exposure among multiple treatments at the same site and among different sites in the same and in different patients.
* Determine the cumulative response achieved at the completion of treatment in these patients.
* Determine the number of sessions required to complete treatment in these patients.
* Correlate ETR with incremental treatment response in patients treated with this regimen.

OUTLINE: This is a randomized study. Patients' individual lesions are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive a short duration of topical aminolevulinic acid (ALA) on the lesion and surrounding normal skin. The lesion is then illuminated with red light for up to 30 minutes.
* Arm II: Patients receive a medium duration of ALA followed by light illumination as in arm I.
* Arm III: Patients receive a long duration of ALA followed by light illumination as in arm I.

In all arms, treatment repeats every 2 weeks for up to 12 courses in the absence of unacceptable toxicity or progressive (systemic) disease.

Additional patients are accrued to a treatment arm if at least 2 of 3 patients on that arm experience 25% cumulative clinical response.

Patients are followed at 1, 3, and 6 months and then every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 4-10 patients will be accrued for this study within 5-7 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* One of the following histologically confirmed diagnoses:

  * Cutaneous B-cell or T-cell lymphoma confined to the skin

    * No evidence of internal disease other than peripheral adenopathy
  * Early chronic lymphocytic leukemia with cutaneous B-cell infiltrates not requiring systemic therapy
* Stable or slowly progressive disease that is not expected to substantially change during treatment

PATIENT CHARACTERISTICS:

Age

* Not specified

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant or nursing
* No porphyria or known hypersensitivity to porphyrins
* No known photosensitivity diseases

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Concurrent clinically necessary interferon alfa allowed

Chemotherapy

* No concurrent systemic multiagent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No concurrent local radiotherapy to study lesions
* No concurrent whole body radiotherapy

Surgery

* Not specified

Other

* More than 1 month since prior topical therapy to study lesions
* Concurrent topical therapy to non-study lesions allowed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 1999-02; Primary Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Pain grade and epidermal toxic response (ETR)
Feasibility of maintaining a pain grade of 1 or less and an approximate ETR of 2
Maximal irradiance and corresponding exposure
Cumulative response achieved at the completion of treatment
Number of sessions required to complete treatment
Correlation of ETR with incremental treatment response

CONTACTS AND LOCATIONS:
Overall Officials: Allan R. Oseroff, MD, PhD, Study Chair — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States